CLINICAL TRIAL: NCT06467968
Title: GATED-PET Heart Analysis in Patients Having a Gallium-68--DOTATOC PET/CT Exam for Oncology Indication
Brief Title: Heart Analysis in GATED-PET in Patients Having a Gallium-68-DOTATOC PET/CT Exam for Oncology Indication
Acronym: GATEDOTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mathieu PERRIN, MD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022PI008
Record Dates: First submitted 2022-07-07; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Inflammation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Person for whom a 68Ga-DOTATOC PET/CT exam is requested as part of the diagnostic or pre-therapeutic assessment of a neuroendocrine tumor
  Interventions: Other: Cardiac ECG-gated PET imaging will added

INTERVENTIONS:
Other: Cardiac ECG-gated PET imaging will added — Blood sample will be used to measure troponin, BNP and CRP . After 68Ga-DOTATOC PET/CT whole body recording, a cardiac ECG-gated PET imaging will added
  Other Names: blood sample

SUMMARY:
Gallium-68-DOTATOC binds primarily with high affinity to somatostatin subtype 2 (SSTR2) receptors and these somatostatin receptors are also overexpressed on inflammation cells when activated.

The hypothesis is that the GATED mode on a Gallium-68-DOTATOC cardiac recording would be able to highlight abnormalities that could be correlated with the age of the patients and their cardiovascular risk factors.

DETAILED DESCRIPTION:
People with the selection criteria for the study, coming to the nuclear medicine department in order to benefit from a Gallium-68-DOTATOC PET/CT exam as part of a diagnostic or pre-therapeutic assessment of a neuroendocrine tumor will be offer to participate in the study After sign consent, patients were install in a room to have blood drawn for Troponin Ic, BNP and CRP and after Gallium-68-DOTATOC infusion Gallium-68-DOTATOC PET/CT will be recorded and immediately the cardiac record in Gated mode

ELIGIBILITY:
Inclusion Criteria:

Persons who have received complete information on the organization of the research and who have signed the informed consent and:

* Age ≥ 18 years old.
* Having read and understood the information document.
* Affiliated to a social security scheme.

Person for whom a 68Ga-DOTATOC PET/CT exam is requested as part of the diagnostic or pre-therapeutic assessment of a neuroendocrine tumour.

Exclusion Criteria:

Person with

* Hypersensitivity during previous use of 68Ga-DOTATOC
* Impossibility of performing a PET-CT (patient agitated, confused, etc.).
* History of heart disease,
* Severe arrhythmia that does not allow the PET synchronized with the ECG
* Severe renal insufficiency (GFR <30 ml/min/1.73 m2)
* Treated with a somatostatin analogue.
* Cushing's syndrome
* Pregnant woman, likely to be or breastfeeding
* Adult subject to a legal protection measure (guardianship, curators, legal safeguard)
* Person of legal age unable to express their consent
* Person deprived of liberty by a judicial or administrative decision
* Person, subject to psychiatric care under articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
Relationship between the captation of radiotracer and the cardiovascular disease | 1 day
  Measurement of myocardial activity

SECONDARY OUTCOMES:
Relationship between the captation of radiotracer and the troponin value | 1 day
  Correlation between the myocardial activity and the troponin value

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu PERRIN, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Veronique Roch, Vandœuvre-lès-Nancy, France